CLINICAL TRIAL: NCT07336602
Title: Immediate and Sustained Effects of Intensive Neuroproprioceptive Equine-Assisted Physiotherapy in Children With Spinal Muscular Atrophy: A Randomized Crossover Trial
Brief Title: Neuroproprioceptive Equine-Assisted Physiotherapy for Spinal Muscular Atrophy
Acronym: NEUROEQUIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, proffesor, Charles University, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4424; GAUK 4424/2024 (Other Grant/Funding Number: Charles University); SVV 260533/SVV/2024 (Other Grant/Funding Number: Charles University); Cooperatio Neurosciences (Other Grant/Funding Number: Charles University)
Record Dates: First submitted 2025-11-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: Muscular atrophy, Spinal; Genetic Therapy; Equine-Assisted Therapy; Child; Pediatrics; Physical Therapy Modalities; RNA, Long Noncoding; Neuro-proprioceptive Principles
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Participants first receive NEUROEQUIP-SMA (Equine-Assisted Physiotherapy Based on Neuro-proprioceptive Facilitation and Inhibition) for six consecutive days, followed by a washout period of 6 weeks to 3 months, and then Standard Individual Outpatient Physiotherapy Based on Neuro-proprioceptive Facilitation and Inhibition (SMA-SOC-N) for six consecutive days. Each phase includes standardized Therapeutic Grooming.
  Interventions: Behavioral: Equine-Assisted Physiotherapy based on Neuro-proprioceptive "Facilitation and Inhibition"; Behavioral: Standard Individual Outpatient Physiotherapy Based on Neuro-proprioceptive Facilitation and Inhibition; Behavioral: Therapeutic grooming
- Sequence B (Experimental): Participants first undergo six days of standard individual outpatient physiotherapy based on neuro-proprioceptive facilitation and inhibition (SMA-SOC-N), followed by a washout period of 6-12 weeks, and then six days of equine-assisted physiotherapy based on neuro-proprioceptive facilitation and inhibition (NEUROEQUIP-SMA). Each phase includes a standardized therapeutic grooming component.
  Interventions: Behavioral: Equine-Assisted Physiotherapy based on Neuro-proprioceptive "Facilitation and Inhibition"; Behavioral: Standard Individual Outpatient Physiotherapy Based on Neuro-proprioceptive Facilitation and Inhibition; Behavioral: Therapeutic grooming

INTERVENTIONS:
Behavioral: Equine-Assisted Physiotherapy based on Neuro-proprioceptive "Facilitation and Inhibition" — Equine-assisted physiotherapy applying the principles of neuro-proprioceptive facilitation and inhibition. Conducted twice daily for 15 minutes over six consecutive days under the supervision of a certified physiotherapist and a trained horse leader. The intervention utilizes the horse's rhythmic, three-dimensional movement to generate dynamic proprioceptive, vestibular, and tactile stimuli that activate physiological postural reactions and coordinated muscle chains. The goal is to improve trunk stability, breathing control, movement symmetry, and functional motor coordination in children with spinal muscular atrophy. The therapy is delivered in a controlled equine environment, using manual facilitation and specific body positioning to modulate neuronal excitability and enhance neuromuscular function.
  Other Names: NEUROEQUIP-SMA
Behavioral: Standard Individual Outpatient Physiotherapy Based on Neuro-proprioceptive Facilitation and Inhibition — Standardized outpatient physiotherapy program based on neuro-proprioceptive facilitation and inhibition, performed once daily for 30 minutes over six consecutive days. Delivered by an experienced physiotherapist in a clinical setting, the intervention includes active and assisted movement exercises, breathing techniques, stretching, postural correction, and positioning strategies to prevent contractures, maintain range of motion, and support trunk and respiratory control. The therapy applies targeted afferent stimuli to modulate motoneuron excitability and improve voluntary activation of motor units. The approach follows international standards of SMA rehabilitation, focusing on optimizing postural alignment, movement efficiency, and overall motor performance.
  Other Names: SMA-SOC-N
Behavioral: Therapeutic grooming — Structured horse-care activity included in both treatment periods to control for psychosocial and environmental effects of horse interaction. Conducted once daily for approximately 20 minutes under therapist supervision, therapeutic grooming involves guided brushing, tactile contact, and communication with the horse in a safe and supportive setting. The activity promotes sensory integration, body awareness, and emotional regulation, while preparing the child for subsequent equine-assisted sessions. Although not a primary therapeutic modality, it standardizes the environmental exposure across study arms and supports comfort, motivation, and engagement in children participating in physiotherapeutic interventions.

SUMMARY:
This study investigates whether Equine-Assisted Physiotherapy based on Neuro-proprioceptive "Facilitation and Inhibition" (NEUROEQUIP-SMA) can improve movement, posture, breathing, and quality of life in children with spinal muscular atrophy (SMA). This therapy uses the horse's rhythmic movement together with targeted sensory and manual stimulation to trigger natural motor reactions starting from the pelvis, lower the threshold for muscle activation, and support coordinated motor patterns. The study compares this method with standard individual physiotherapy based on the same neuro-proprioceptive facilitation and inhibition principles, but performed without the horse. Twenty children aged 2 to 9 years will receive both therapies in two separate 6-day blocks, in random order (crossover design). The researchers will assess muscle fatigue, coordination, breathing function, movement quality and quantity, quality of life, and changes in selected blood biomarkers. The results may help develop better rehabilitation strategies for children with SMA who are receiving modern pharmacological or gene therapy.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is an autosomal recessive neuromuscular disorder caused by deletions or mutations of the SMN1 gene with retention of its paralog SMN2. Despite recent advances in disease-modifying treatments, SMA remains the leading genetic cause of infant mortality and continues to require multidisciplinary supportive care to achieve optimal outcomes. Physiotherapy is an integral part of this care, helping to maintain mobility, prevent contractures, and enhance quality of life.

Historically, physical activity was discouraged in SMA because of concerns that exercise might accelerate motor-neuron degeneration. Subsequent evidence has shown that inactivity contributes to weakness and fatigue, whereas appropriately dosed physical therapy improves postural control, endurance, and respiratory function. Modern rehabilitation therefore emphasizes functional mobility, balance training, and gait rehabilitation. Experimental studies have also demonstrated that specific exercise parameters can activate neuroprotective mechanisms independent of SMN protein expression, suggesting that motor-unit activation itself may support neuronal health.

Building on these findings, the present study introduces Equine-Assisted Physiotherapy Based on Neuro-proprioceptive "Facilitation and Inhibition" (NEUROEQUIP-SMA)-an innovative physiotherapeutic approach designed for children with SMA. This method combines the dynamic multisensory input of equine movement with the principles of neuroproprioceptive facilitation and inhibition, in which appropriate afferent stimuli modulate interneuronal excitability to optimize transmission within motor pathways. The technique aims to lower the excitability threshold of motor neurons so that impulses from the central nervous system can effectively induce muscular activation. Similar neurofacilitation strategies are routinely used in Czech neurorehabilitation for patients after stroke or with multiple sclerosis, but their potential in SMA has not yet been systematically studied.

The NEUROEQUIP-SMA method is compared with a standard physiotherapy program based on neuroproprioceptive facilitation and inhibition principles delivered in an outpatient setting. Both approaches target postural alignment, trunk stability, and functional motor control. The equine-assisted modality is expected to further enhance outcomes by promoting rhythmic pelvic activation, symmetric weight shifting, coordinated engagement of weakened muscle chains, and improved respiratory patterning through the horse's cyclic movement.

The study uses a randomized crossover design to evaluate short-term effects after an intensive six-day program. Primary outcomes include changes in motor function, postural control, and respiratory parameters, complemented by surface electromyography to monitor muscle fatigue. Secondary measures address quality of life, psychomotor development, and parent-reported well-being.

As an exploratory molecular component, peripheral blood will be analyzed for selected long non-coding RNAs (lncRNAs) such as SMN-AS1, MALAT1, PARTICLE, MEG3, NEAT1, H19, and GAS5. These transcripts are involved in motor-neuron development and chromatin regulation through PRC2-associated mechanisms. Their expression changes may serve as potential biomarkers reflecting neurophysiological effects of intensive physiotherapy in SMA.

The study was reviewed and approved by the Ethics Committee of the Third Faculty of Medicine, Charles University, Prague, Czech Republic. The intervention is short-lasting, low-risk, and non-pharmacological; therefore, a formal Data Monitoring Committee was not required. The findings are expected to contribute to evidence-based recommendations for physiotherapeutic management of SMA and to provide insight into the molecular correlates of motor-function improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 9 years
* Clinical diagnosis of spinal muscular atrophy (SMA) type I, II, or III
* Stable health condition for at least 6 months prior to enrollment
* Ability to participate in the study procedures
* Written informed consent provided by a parent or legal guardian

Exclusion Criteria:

* Hip dislocation
* Known allergy to horses or the stable environment
* Severe fear of horses that would prevent participation in equine-assisted physiotherapy

Any other medical condition that, in the investigator's opinion, would interfere with safe participation in the study

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  A clinical assessment tool used to evaluate motor function in infants with neuromuscular disorders measures their ability to perform specific movements and assesses the severity of motor impairments. Measurements are recorded during the test and are later evaluated by two independent physiotherapists. Scores range from 0 to 64, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Change in Relative Expression of Selected lncRNAs | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of 28 days from the end of the intervention.
  Relative expression of a predefined panel of long non-coding RNAs (lncRNAs) in peripheral blood, measured by quantitative PCR and normalized to reference genes. For reporting purposes, the mean fold change across the predefined lncRNA panel will be calculated and reported as a single outcome value.
Change in Median Frequency of Surface EMG Signal | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  Median frequency of the surface electromyography (sEMG) signal recorded from the external oblique abdominal muscle during a standardized repetitive movement task. Lower median frequency values over repeated contractions indicate improved muscle efficiency and reduced fatigue.
The Trunk Control Measurement Scale (TCMS) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  The Trunk Control Measurement Scale (TCMS) is a clinical assessment tool that evaluates trunk control during static and dynamic sitting balance tasks. It measures selective movement control in the trunk and coordination between upper and lower body segments. Although validated primarily in children with cerebral palsy, it is also used to assess postural control in children with other neuromotor disorders such as SMA. The total score ranges from 0 to 58, with higher scores indicating better trunk control.
The Segmental Assessment of Trunk Control (SATCo) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  The Segmental Assessment of Trunk Control (SATCo) is a standardized test designed to identify the highest level of segmental trunk control in sitting. It assesses static, active, and reactive control at seven levels of trunk support. Although originally developed for children with cerebral palsy, it has been used in other pediatric neuromotor populations to evaluate trunk stability and postural development. Scores range from 0 to 20, with higher scores indicating better trunk control.
Motor Function Measure-20 (MFM-20) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  The Motor Function Measure-20 (MFM-20) is a validated quantitative scale assessing motor skills in children with neuromuscular disorders aged 2-7 years. It contains 20 items covering standing, transfer, axial and proximal motor functions, and distal motor control. The total score is expressed as a percentage of the maximum possible score, with higher scores indicating better motor performance. The MFM-20 has been validated in SMA and Duchenne muscular dystrophy and is sensitive to changes over time. Scores range from 0 to 100%, with higher scores indicating better motor function.
The Functional Reach Test (FRT) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  The Functional Reach Test (FRT) is a simple, validated measure of dynamic sitting or standing balance that evaluates the maximal distance an individual can reach forward beyond arm's length while maintaining a fixed base of support. It is a reliable indicator of trunk stability and balance control in children with various neuromotor conditions, including SMA. Longer reach distances indicate better dynamic postural control and balance performance.
The Selective Control of Lower Extremities (SCALE) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  The SCALE test is a standardized clinical test used to assess selective voluntary motor control in the lower extremities. It assesses the ability to isolate joint movements during five tasks for each lower extremity. Each joint movement is scored from 0 to 2, and a higher total score indicates better selective motor control.
Change in Angle of Trunk Rotation | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  Angle of trunk rotation (ATR) measured during standardized forward bending in the sitting position. The mean ATR value will be calculated from repeated measurements and reported as a single outcome value.
Change in Forced Expiratory Volume in One Second (FEV₁) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  Forced expiratory volume in one second (FEV₁) measured by standard spirometry. Higher values indicate better pulmonary function.
Change in Maximum Displacement of Body Markers | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  Maximum displacement of predefined body markers from their initial position during a standardized reaching task performed in sitting. Greater displacement values indicate improved control of the center of gravity.
Change in Abdominal Breathing Index | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  Abdominal breathing index calculated as the ratio of marker displacement at the lumbar level (L4) to displacement at the thoracic level during deep breathing. Higher values indicate a greater contribution of abdominal breathing.
Change in Duration of Coordinated Trunk and Cervical Spine Movement | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 6-day intervention.
  Duration of coordinated trunk and cervical spine movement during a standardized repetitive upper limb task performed in sitting. Longer durations without compensatory cervical spine extension indicate improved coordination.
Quality of life questionnaire | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of 28 days from the end of the intervention.
  Parents of children with SMA will complete a special questionnaire at the beginning and 28 days after the end of the rehabilitation. The ICF score set, specifically the ICF-based Documentation Form for the category "Children with Cerebral Palsy Brief" (for children under 6 years old), will be used to evaluate the quality of life. A Higher scores indicate better functioning and quality of life.
Pediatric Quality of Life Inventory Generic Core Scales (PedsQL™) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of 28 days from the end of the intervention.
  The assessment tool, designed to evaluate health-related quality of life in children, consists of 23 items across four domains (physical, emotional, social, and school functioning). It is used to monitor longitudinal changes in perceived quality of life and to evaluate the effectiveness of clinical and rehabilitative interventions. Scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Change in Video-Based Motor Function Score | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of 28 days from the end of the intervention.
  Motor function score derived from standardized evaluation of home video recordings by two independent physiotherapists. The score reflects the quality and extent of the child's movement. Scores range from 1 to 21, with higher scores indicating better motor function.
Strengths and Difficulties Questionnaire (SDQ) | Baseline measurement before the start of the 6-day intervention, follow-up measurement after the end of the 28-day intervention.
  The SDQ is a widely used behavioral screening tool assessing psychological attributes across five domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. It is suitable for children aged 2 to 17 years and provides a Total Difficulties Score reflecting overall psychosocial well-being. Although originally validated in the general pediatric population, it has been successfully applied in children with chronic or neuromuscular disorders to assess emotional and social adaptation related to health status. Scores range from 0 to 40, with higher scores indicating greater behavioral and emotional difficulties.
Change in Peak Expiratory Flow (PEF) | Baseline measurement before the start of the 6-day intervention and follow-up measurement after the end of the 6-day intervention.
  Peak expiratory flow (PEF) measured by standard spirometry. Higher values indicate better pulmonary function.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Marikova, master, Principal Investigator — Charles University, Czech Republic
Locations (4):
- Czechia (4):
  - Mirákl Hippotherapy Center, Bohuslavice
  - College of Polytechnics Jihlava, Jihlava
  - Department of Medical Genetics, Third Faculty of Medicine, Charles University, Prague
  - Third Faculty of Medicine, Charles University, Prague

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in publications (after de-identification) may be shared. This includes anonymized outcome data, demographic characteristics, and relevant clinical variables used for statistical analysis. The study involves a short-lasting, low-risk, non-pharmacological intervention; therefore, no Data Monitoring Committee (DMC) is established. After completion of data analysis, de-identified datasets will be available upon reasonable request to the corresponding author. Data will be shared for legitimate scientific purposes, such as meta-analyses and systematic reviews, in compliance with ethical and institutional regulations. The results of the study will also be disseminated through peer-reviewed publications and conference presentations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of data analysis and publication of primary results (expected 2026-2027); data will be available for at least 10 years thereafter.
Access Criteria: De-identified individual participant data (IPD) will be shared only if permitted by the signed informed consent. Identifiable data will remain accessible solely to the study team and will not be shared. Qualified researchers may request access to de-identified IPD for scientific purposes by emailing the corresponding author with a brief proposal and data-use agreement. Data will be transferred securely and handled in compliance with GDPR and institutional policies; recipients must agree not to attempt re-identification.

REFERENCES:
- [Result] Lemke D, Rothwell E, Newcomb TM, Swoboda KJ. Perceptions of equine-assisted activities and therapies by parents and children with spinal muscular atrophy. Pediatr Phys Ther. 2014 Summer;26(2):237-44. doi: 10.1097/PEP.0000000000000027. PMID 24675128
- [Result] Pantera E, Froment P, Vernay D. Does Hippotherapy Improve the Functions in Children with Cerebral Palsy? Systematic Review Based on the International Classification of Functioning. J Integr Complement Med. 2022 Sep;28(9):705-720. doi: 10.1089/jicm.2021.0417. Epub 2022 Jun 7. PMID 35671520
- [Result] Rasova K, Buckova B, Prokopiusova T, Prochazkova M, Angel G, Markova M, Hruskova N, Stetkarova I, Spanhelova S, Mares J, Tintera J, Zach P, Musil V, Hlinka J. A Three-Arm Parallel-group Exploratory Trial documents balance improvement without much evidence of white matter integrity changes in people with multiple sclerosis following two months ambulatory neuroproprioceptive "facilitation and inhibition" physical therapy. Eur J Phys Rehabil Med. 2021 Dec;57(6):889-899. doi: 10.23736/S1973-9087.21.06701-0. Epub 2021 Feb 10. PMID 33565742
- [Result] Trenkle J, Brugman J, Peterson A, Roback K, Krosschell KJ. Filling the gaps in knowledge translation: Physical therapy recommendations for individuals with spinal muscular atrophy compared to standard of care guidelines. Neuromuscul Disord. 2021 May;31(5):397-408. doi: 10.1016/j.nmd.2021.02.011. Epub 2021 Feb 16. PMID 33741230
- [Result] Mercuri E, Sumner CJ, Muntoni F, Darras BT, Finkel RS. Spinal muscular atrophy. Nat Rev Dis Primers. 2022 Aug 4;8(1):52. doi: 10.1038/s41572-022-00380-8. PMID 35927425
- [Result] Voight S, Arya K. Considerations for Treatment in Clinical Care of Spinal Muscular Atrophy Patients. Children (Basel). 2024 Apr 20;11(4):495. doi: 10.3390/children11040495. PMID 38671712
- [Result] Shin HI. Rehabilitation Strategies for Patients With Spinal Muscular Atrophy in the Era of Disease-Modifying Therapy. Ann Rehabil Med. 2024 Aug;48(4):229-238. doi: 10.5535/arm.240046. Epub 2024 Aug 30. PMID 39210748
- See also: Official website of the coordinating institution and study sponsor. — https://www.lf3.cuni.cz/
- See also: Clinical site for equine-assisted physiotherapy (NEUROEQUIP-SMA). — https://www.chmirakl.cz/
- See also: Reference for the ICF Core Set used in functional assessment. — https://www.icf-research-branch.org/
- See also: Information about the university grant funding the study. — https://cuni.cz/UK-9291.html